CLINICAL TRIAL: NCT04744337
Title: Temporomandibular Joint Adaptations After Fixed Orthodontic Therapy in Cases Already Treated With Twin Block Appliance
Brief Title: TMJ Adaptations by Orthodontic Treatment in Adolescent Females With Angle's Class II Division 2 Malocclusion: MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Preeti Nain
Record Dates: First submitted 2018-09-15; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Class II Division 2 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orthodontic treatment (Other): fixed orthodontic treatment in adolescent females initially treated with removable functional appliance for skeletal class II, Angle's class II division 2 malocclusion.
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Procedure: orthodontic treatment — fixed orthodontic treatment in adolescent females initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion.
  Other Names: fixed mechanotherapy

SUMMARY:
The aim of this study is to document the changes brought about in the internal anatomic relationships of the TMJ complex,positional changes of glenoid fossa with respect to adjacent cranial structures after completion of fixed orthodontic treatment in adolescent females initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 Malocclusion.

DETAILED DESCRIPTION:
Angle's class II division 2 malocclusion is subtype of Angle's class II malocclusion with unique facial, dental and craniofacial features which differentiate it from other malocclusions so much that it has been said to be a syndrome itself. Its frequency lies between 1.5 and 5% of all malocclusions found in a white western population. Hypertrophic masticatory muscles as documented in class II division 2 are directed in more anterior direction leading to increased magnitude of occlusal forces and hence increased TMJ loading. TMJ morphology depends, to an extent on occlusal loads acting on it, so class II division 2 malocclusion patients are expected to have specific TMJ complex morphology. Condyle position changes from anterior to posterior with age in class II division 2 cases. The use of functional orthopedic appliances to correct Class II malocclusions associated with retrognathic mandibles is indicated for the first phase of orthodontic treatment. A second phase of treatment is undertaken with fixed orthodontic appliances to obtain occlusal refinement. Although various investigations have shown the efficiency of this method of treatment, the mechanism by which the temporomandibular joint (TMJ) responds to the treatment is controversial.

Various techniques have been used to image the TMJ which include Magnetic Resonance Imaging (MRI), Cephalograms, Orthopantomograms , Tomograms , Bone scintigraphy with radiologic markers like 99mTc-MDP, Arthroscopy and Arthrography , CT scanning, Cone Beam Computed Tomography (CBCT).

Magnetic Resonance Imaging (MRI), a multiplanar imaging technique, has the advantage of giving an accurate assessment of both the bony and the soft tissues. This technique is believed to be non-invasive, radiation free and gives more superior contrast resolution than any other imaging modality. MRI is considered the imaging modality of choice for assessment of internal derangements of the temporomandibular joint. According to Akar et al "Bony structures and especially soft tissues of the TMJ can be examined by means of MRI and the relations of the tissues with each other can be evaluated." MRI studies have been done on fixed functional appliances which show significant displacement of condyle during treatment but later condyles returned to pre treatment positions at the end of fixed functional appliance treatment. Results documented in fixed functional appliance may not be same in removable appliances. Effects of removable functional appliances on the condyle-glenoid fossa (C-GF) complex have been studied with respect to the Frankel, Activator, Twin block and Bionator appliances. Franco et al found that Frankel therapy resulted in a 'more normal' articular disc morphology. Arat et al. concluded that disc positions were insignificant after 6 months of Activator therapy Chintakanon et al. concluded that Twin Block therapy had neither positive nor negative effects on disc position, and there was little evidence that the disc was recaptured. They also noted anterior positioning of the condylar head (CH) in the glenoid fossa after 6 months of Twin Block therapy. It should be noted that all of above studies are limited to the phase of removable functional appliance therapy only in Class II division 1 and no MRI study has attempted to evaluate the changes in the position of the Condyle-Glenoid Fossa (C-GF) complex treated with removable functional appliance therapy, followed by fixed orthodontic treatment in Class II division 2 malocclusion.

Aidar et al have studied changes in temporomandibular joint disc position and form following Herbst and fixed orthodontic treatment and found that at the end of the bi-phasic treatment the position and form of the initial articular discs were maintained. Kinzinger, et al. studied the effects of fixed orthodontic treatment in the case of skeletal class II on the position of the articular disc and condyle using MRI on 20 subjects and concluded that treatment did not alter the position of articular disc and even noticed an improvement in the anterior disc displacement in 8 joints out of 40. No studies have been done on bi-phasic treatment of skeletal class II, Angle's class II division 2 involving removable functional appliances in the first phase followed by fixed orthodontic treatment in second phase.

Therefore, the aim of this study is to document the changes brought about in the internal anatomic relationships of the TMJ complex , positional changes of glenoid fossa with respect to adjacent cranial structures after completion of fixed orthodontic treatment in adolescent females initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion,

MATERIALS AND METHODS

It is a longitudinal clinical trial to evaluate TMJ disc-condyle-fossa relationship using MRI scan following bi-phasic therapy in skeletal Class II, Angle's class II division 2 malocclusion in adolescent females.

The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopedics, PGIDS, in association with the Department of Radiology, PGIMS, and Department of Oral Radiology, PGIDS, Pt B. D. Sharma University of Health Sciences, Rohtak.

Ethical clearance- The study will be carried out in humans after the institutional approval obtained from ethical committee.

Source of Data The study sample will consist of the subjects from the Department of Orthodontics and Dentofacial Orthopedics, PGIDS , who will be successfully completing the prefunctional and functional appliance therapy for correction of skeletal class II, Angle's class II division 2 malocclusion and will be ready for fixed orthodontic treatment for final finishing and detailing of occlusion

INFORMED CONSENT OF THE PATIENT

A valid, bilingual informed written consent of the patient or parent/guardian will be obtained from the patient before registering the patient in this clinical study. Patients will be informed of all the theoretical risks and benefits of the interventions under test.

Intervention and design of study The study sample will consist of those 14 adolescent females who had been treated initially with pre functional and functional appliance therapy for skeletal Class II, Angle's class II division 2 malocclusion and had following MRI scans done during the treatment

Stage- A (pre-treatment), Stage- B (after pre-functional therapy) Stage- C (After completion of Functional Appliance Therapy) These patients will be further treated with fixed orthodontic treatment for final finishing and detailing and an MRI will be taken after debonding of fixed orthodontic appliance (stage D). MRI scans thus obtained will be evaluated for documenting changes in the morphology and anatomic positions of condylar head, articular disc and glenoid fossa and will be traced for the various angular and linear metric measurements MRI scans of the TMJ will be obtained with a 1.5/3 Tesla Philips Intera Nova Gradient (Netherlands) scanner equipped with Sense Head 6 channel coil for simultaneous imaging of right and left joints. Sagittal images will be taken perpendicular to the long axis of the condylar head and the coronal images will be taken parallel to the long axis of the condylar head. The images will be recorded in maximum intercuspation after debonding of fixed orthodontic appliance. The MRI protocol will include PD TSE (Turbo Spin Echo) sequence (TR 1500/ TE 30/ FoV 150x150 mm) T1 spin echo sequences (TR 450⁄TE 15⁄FoV 160x160 mm) and T2 TSE sequence (TR 2424⁄ TE 100⁄FoV 160x160 mm).

FIXED MECHANOTHERAPY TREATMENT PHASE

The sample will be having cases in class I/ superclass I molar relation and lateral open bite may be present in premolar regions after the completion of functional phase. The final fixed orthodontic phase will be taken up for the final finishing and detailing of the occlusion after the retentive phase of functional appliance therapy is completed. It involves banding and bonding of both upper and lower arches with MBT 0.022" appliance. Progressive wire sequences to be used are 0.014" NiTi, 0.016" NiTi, 0.018" NiTi, 0.017" x 0.025" NiTi, 0.019"x 0.025" NiTi, , 0.019"x 0.025" S.S., 0.014" S.S. Once stainless steel archwires are in place, class II elastics may be prescribed to the patient to prevent relapse of class I molar relation achieved. Cases are to be finished in class I molar intercuspation with normal overjet and overbite. Appliance will be debonded and final MRI (stage D) will taken for all the patients. Hawley's retainer with anterior bite plane will serve for retention of achieved results

Evaluation of MRI stages

This will be done with the help of following parameters:

ANGULAR AND LINEAR MEASUREMENTS The eminence angle and the sagittal disc position measured in relation to two reference lines: the posterior condylar line (PC line) and the Frankfurt Horizontal plane (FH Plane). The PC line to be drawn directly on the MRI scan, while the FH plane transferred from the lateral cephalogram to the MRI scan, according to the method given by Nebbe et al.

Transfer of FH plane Determination of long axis of the condyle will be done by two step circle center method by Nebbe et al.

ANGULAR MEASUREMENTS 1-2) The eminence angle and the coronal disc position will be evaluated by the method described by Chintakanon et al.

3) The sagittal disc position will be evaluated using PC line and FH plane as described by Chintakanon et al.

4) Sagittal condylar concentricity will be evaluated using the method described by Pullinger et al.

5) The glenoid fossa angle will be measured on the sagittal films as the angle between the tangents to the anterior and posterior slopes of the glenoid fossa.

LINEAR MEASUREMENTS 6) Condyle and glenoid fossa displacements: The position of the glenoid fossa, and that of the condyle, will be evaluated with respect to the centre of the external auditory meatus (c-EAM). by marking one point at the centre of condyle (c-CH) and the linear distance of the c-CH from the c-EAM will be evaluated as the shortest distance from the constructed FH perpendicular.

7) Distance between c-PGS (crest of the post-glenoid spine ) & c-EAM : One point will be marked at the crest of the post-glenoid spine (c-PGS) and the linear distance of the c-PGS from the c-EAM will be evaluated as the shortest distance from the constructed FH perpendicular.

8) Superior joint space will be measured from the shortest distance between the most superior point of the condyle and the most superior point of the mandibular fossa.

Statistical analysis The final data recorded will be processed by standard statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Cases with moderate skeletal Class II bases with mandibular retrognathia, Angle's Class II division 2 malocclusion treated initially with prefunctional and functional appliance therapy in their active growth period and will be ready for fixed orthodontic treatment and have had MRI done at following stages:

  1. Stage- A (pre-treatment)
  2. Stage- B (after pre-functional therapy)
  3. Stage-C (After completion of functional appliance therapy)

Exclusion Criteria:

* 1.Patients with any internal derangement or pathology of TMJ. 2.History of systemic diseases affecting bone metabolism. 3.Growth abnormality. 4.Bleeding disorders. 5. Patients with facial asymmetry.

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — females
Enrollment: 14 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
MRI comparisons for TMJ adaptations in adolescent females | 12 months
  TMJ adaptations with the help of various angular and linear measurements in adolescent females before and after fixed orthodontic therapy who were initially treated with functional appliance therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Nain, MDS student, Principal Investigator — PGIDS Rohtak, Haryana
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No
The aim of this study is to document the changes brought about in the internal anatomic relationships of the TMJ complex, positional changes of glenoid fossa with respect to adjacent cranial structures after completion of fixed orthodontic treatment in adolescent females initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion.